CLINICAL TRIAL: NCT07013838
Title: Comparison of Deucravacitinib and Adalimumab for the Treatment of Relapsed Takayasu's Arteritis: The TYK-TAK Trial
Brief Title: The Efficacy and Safety of Deucravacitinib in Takayasu's Arteritis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese SLE Treatment And Research Group (Other)
Responsible Party: Principal Investigator, Xinping Tian, Professor of Medicine, Chinese SLE Treatment And Research Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TYK2-TAK-01
Record Dates: First submitted 2025-05-25; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Takayasu Arteritis (TAK)
Keywords: Deucravacitinib; Adalimumab; Relapsed; Efficacy; Safety; Takayasu arteritis
MeSH Terms: conditions — Takayasu Arteritis; Recurrence | interventions — deucravacitinib; Adalimumab

STUDY DESIGN:
Intervention Model Description: prospective, single-center, randomized, open-label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deucravacitinib treatment group (Experimental): Patients randomly assigned to the deucravacitinib treatment group are required to take the deucravacitinib tablets 6mg orally once daily on an empty stomach or after a meal during D1-D168, and orally take the study drug deucravacitinib with warm water. It is forbidden to drink water from 1 h before administration to 1 h after administration (except for administration of water) and fasting within 1 h after administration. Continuous treatment for 168 days or subject discontinuation criteria were met. The time of dose administration is called "0" hour. Subjects who miss a study medication on one day are not allowed to take a supplement to compensate but should take the next dose.
  Interventions: Drug: Deucravacitinib
- Adalimumab treatment group (Active Comparator): Participants assigned to the adalimumab treatment group receive adalimumab 40mg by subcutaneous injection every 2 weeks during D1-D168. Adalimumab is administered for 24 weeks unless the discontinuation criteria are met.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Deucravacitinib — Deucravacitinib is a new, oral, selective, allosteric inhibitor of TYK2. It was first approved in the United States on 09-Sep-2022 for the treatment of adults with moderate-to-severe plaque psoriasis who are candidates for systemic therapy or phototherapy.
  Arms: Deucravacitinib treatment group
Drug: Adalimumab — TNFα inhibitors have already been used in TAK treatment. Several retrospective studies have demonstrated the treatment effects of these agents in patients with TAK, including disease remission, GC tapering and vascular inflammation control. According to the ACR and EULAR guidelines, TNFis are recommended to be considered in cases of relapsing or refractory TAK. These agents (including adalimumab) are the most frequently analyzed therapeutic modalities in recent studies of TAK.
  Arms: Adalimumab treatment group

SUMMARY:
This is a 24-week, single-center, randomized, open-label trial conducted by Peking Union Medical College Hospital. The aim of this study is to assess the efficacy and safety of deucravacitinib in adult patients with relapsing TAK in comparison to patients treated with TNF inhibitor (TNFi), the most well-recognized therapeutic choice of non-glucocorticoid immunosuppressive for patients with relapsed or refractory TAK.

DETAILED DESCRIPTION:
Background:

The majority of patients with TAK experience relapses, and some patients fail to respond adequately to current medications used for treatment of TAK. There is an urgent unmet need to identify novel therapies to effectively treat TAK. Th-17 and Th-1 cells, and their related cytokines IL-12, IL-23, IL-17, and type I interferon have all been reported to play a role in the pathogenesis of TAK. Tyrosine kinase 2 (TYK2) mediates signaling transduction between these key cytokines and immune cells. Therefore, blocking TYK2 signaling may downregulate potential pathogenic pathways in TAK, and may be a therapeutic alternative. No study has investigated the effectiveness of agents targeting TYK2 in the treatment of TAK so far. In the present study, we aim to investigate whether deucravacitinib, an oral, selective, allosteric inhibitor of TYK2, is effective and safe for patients with relapsed TAK.

Objectives:

To assess the efficacy and safety of deucravacitinib in adult patients with relapsing TAK in comparison to patients treated with TNF inhibitor (TNFi), the most well-recognized therapeutic choice of non-glucocorticoid immunosuppressive for patients with relapsed or refractory TAK.

Overall Design:

This is a 24-week, single-center, randomized, open-label trial conducted by Peking Union Medical College Hospital. Patients enrolled into the study are randomly assigned (in a 1:1 ratio, 25 patients in each group) to receive deucravacitinib or adalimumab (a TNFi). Patients are followed for efficacy and safety at month 1, month 3, and month 6. Adverse events/Serious adverse events are assessed and recorded at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible to be included in the study only if all of the following criteria apply:

  1. Signed Written Informed Consent

     1. Participants fully understand the purpose, nature, method, and possible adverse reactions of the study, willing to consent to the trial and follow study protocol and sign informed consent.
     2. Participants must have signed an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved written informed consent form (ICF) in accordance with regulatory, local, and institutional guidelines. This ICF must be obtained before performing any protocol related procedures that are not part of normal patient care.
  2. Type of Participant and Target Disease Characteristics

     1. Adult patients (aged 18 or older) fulfilling the 2022 ACR/EULAR classification criteria for TAK.
     2. Persistence of active disease or relapse despite treatment with GCs combined with a conventional synthetic or biologics immunosuppressive agent other than TNFi.
     3. Active vasculitis by reader interpretation of FDG-PET at enrollment (by the same reader).
  3. Reproductive Status The investigator or designee shall counsel women of childbearing potential (WOCBP) and male participants who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy.

WOCBP must have a negative highly sensitive specify: urine or serum as required by local regulations pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to the start of study intervention.

A female is eligible to participate if she is not pregnant or breastfeeding and at least 1 of the following conditions applies:

Is not a WOCBP OR Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of < 1% per year) during the intervention period and for at least 5 half-lives after product administration and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction for the same period.

WOCBP and male participants who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception.

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:

  1. Medical Conditions

     1. Severe disease from TAK for which urgent treatment with interventional procedures or bypass surgery is considered necessary
     2. Critical organ involvement of TAK, such as myocardial or coronary artery involvement, or cerebral ischemia
     3. Active hepatitis B or C virus infection, active tuberculosis infection
     4. Malignancy in the past 5 years (with the exception of fully excised non-melanoma skin cancer or cervical carcinoma in situ)
  2. Physical and Laboratory Test Findings

     1. Serum liver enzyme tests 3 times higher than the upper limits of normal range
     2. Estimated glomerular filtration rate ≤ 30 ml/minute
  3. Other Exclusion Criteria

     1. Females who are pregnant
     2. Ever treated with TNFi (including adalimumab) and discontinued due to inadequate response or intolerance.
     3. Any other sound medical, psychiatric, and/or social reason as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate at week 24 | Week 24
  * Overall response is defined as the combination of both complete and partial responses.
  * Complete (treatment) response is defined as the absence or complete resolution of clinical signs and symptoms of active TAK and a patient achieving all of the following:
    1. ESR <20mm/hour;
    2. CRP <10mg/L;
    3. No progression of vessel damage in Doppler ultrasonography or CTA, including no new or worsening mural thickness, or stenosis or dilatation;
    4. Dose of GC <15 mg/day prednisone (or equivalent dosage of other GCs).
  * Partial (treatment) response is defined as the absence or complete resolution of clinical signs and symptoms of active TAK and:
    1. ESR <40mm/hour or decrease by 50% compared to the baseline value;
    2. CRP <20mg/L or decrease by 50% compared to the baseline value;
    3. fulfilling the other two criteria of complete response.
  * The absence or complete resolution of clinical signs and symptoms of active TAK is a pre-required criterion for both complete and partial

SECONDARY OUTCOMES:
Time to clinical remission | from inclusion to the end of the study, 24 weeks in total
  time from the baseline to achieve clinical remission
Disease recurrence after achieving clinical remission | from inclusion to the end of the study, 24 weeks in total
  recurrence rate after achieving clinical remission
Time to disease recurrence | from inclusion to the end of the study, 24 weeks in total
  time from clinical remission to disease recurrence
Changes in erythrocyte sedimentation rate (ESR) | week 4, 12 and 24
  Erythrocyte sedimentation rate (ESR) is an indicator of systemic inflammation, will be reported in mm/h.
Changes in serum C reactive protein (CRP) | week 4, 12 and 24
  serum C reactive protein (CRP) is an indicator of systemic inflammation, will be reported in mg/L
Changes in vascular ultrasonography | from baseline to weeks 12 and 24
  Vascular Doppler ultrasonography of the carotid arteries, subclavian arteries and abdominal aorta
Changes in PET/CT scans | from the baseline to week 24
  PET-CT, including 18F-FDG PET/CT and 68Ga-FAPI PET/CT are performed at baseline and at the end of the study to assess the status of arterial inflammation and fibrosis.
Change in level of cytokines | week 4, 12 and 24
  A cytokine panel are used to evaluate serum levels of cytokines in involved signaling pathways.

CONTACTS AND LOCATIONS:
Overall Officials: Xinping Tian, MD, Principal Investigator — Peking Unione Mdecial College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
only patient's clincial information could be released to public

REFERENCES:
- [Background] Le AM, Puig L, Torres T. Deucravacitinib for the Treatment of Psoriatic Disease. Am J Clin Dermatol. 2022 Nov;23(6):813-822. doi: 10.1007/s40257-022-00720-0. Epub 2022 Aug 12. PMID 35960487